CLINICAL TRIAL: NCT00190658
Title: Safety and Efficacy of Humatrope in Pediatric Patients With Genetic Short Stature (SHOX Gene Defect)
Brief Title: Somatropin Treatment in Patients With SHOX Deficiency and Turner Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2704; B9R-MC-GDFN
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-12-20 (Estimated); Status verified 2010-12

CONDITIONS: Failure to Thrive
MeSH Terms: conditions — Failure to Thrive | interventions — Human Growth Hormone; WW Domain-Containing Oxidoreductase

INTERVENTIONS:
Drug: Somatropin (rDNA origin) for injection

SUMMARY:
This clinical trial will compare the mean first year height velocity of somatropin-treated prepubertal patients with SHOX deficiency with the height velocity of a control group of untreated prepubertal patients with SHOX deficiency. Both groups will be compared to a somatropin-treated group of girls with Turner syndrome. After the second year patients in the control group have the option to receive treatment as well. All patients will optionally be treated until they achieved adult height.

ELIGIBILITY:
Inclusion Criteria:

* Turner Syndrome or SHOX disorder
* SHOX: bone age greater than 10 years for boys, greater than 8 years for girls, Turner: bone age greater than 9 years
* Height below 3rd percentile or height below 10th percentile and growth velocity below 25th percentile
* Prepubertal: For girls, Tanner stage 1, for boys Tanner stage 1 and testicular volume no more than 2 mL

Exclusion Criteria:

* GH deficiency or known insensitivity
* Evidence of tumor activity
* Diabetes mellitus or history of impaired glucose tolerance
* Any severe illness known to interfere growth

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75
Dates: Start 2000-02; Primary Completion 2004-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Comparison of first year height velocity of somatropin-treated versus non-treated patients with SHOX deficiency.

SECONDARY OUTCOMES:
Comparison of second year height velocity of somatropin-treated versus non-treated patients with SHOX deficiency.
Non inferiority to somatropin treated patients with Turner syndrome
Adult height of treated patients

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Chair — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com